CLINICAL TRIAL: NCT00779129
Title: Phase II Trial of Caelyx and Cyclophosphamide in Metastatic Breast Cancer
Brief Title: A Study to Evaluate Safety and Efficacy of Caelyx in Combination With Cyclophosphamide in the Treatment of Metastatic Breast Cancer (P02948)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02948
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Caelyx 35 mg/m2 and Cyclophosphamide 600 mg/m2
  Interventions: Drug: Pegylated Lyposomal Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pegylated Lyposomal Doxorubicin — Caelyx 35 mg/m2 intravenously, on Day 1, every 3 weeks, during 6 cycles. Patients still achieving clinical benefit after a total of 6 cycles may continue therapy.
  Other Names: SCH 200746
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2, intravenously, on Day 1, every 6 weeks, during 6 cycles (concomitantly with Caelyx). Patients still achieving clinical benefit after a total of 6 cycles may continue therapy.

SUMMARY:
Women with metastatic breast cancer are usually treated with anthracyclines (ie, doxorubicin or epirubicin) but cardiac toxicity limits their use. The aim of this study is to evaluate the safety and efficacy of Caelyx in combination with cyclophosphamide in women with metastatic breast cancer who have received adjuvant anthracyclines with or without a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged >=18 years.
* Subject must have histologic diagnosis of breast carcinoma.
* Subject must have documented measurable metastatic breast cancer by appropriate radiologic imaging.
* Subject must have previous anthracyclin-based adjuvant regimen and disease-free status for at least one year following the completion of adjuvant therapy.
* Subject must have ECOG performance status 0, 1, or 2.
* Subject must have life expectancy > 6 months
* Subject must have left ventricular ejection fraction >=55% as determined by MUGA scan.
* Subject must have normal organ function, except if abnormal due to tumor involvement:

  * Adequate bone marrow function (platelets >=100 X 10^9/L, hemoglobin >=90 g/L, Neutrophils >=1.5 X 10^9/L)
  * Adequate renal function (serum creatinine < 2 X the upper limit of normal (ULN)
  * Adequate liver function (bilirubin < 2 times ULN, AST or ALT < 2 times ULN in the absence of liver metastasis, AST or ALT < 5 times ULN in the presence of liver metastasis.
* Women of childbearing potential must be using adequate contraception and have a negative pregnancy test at the time of enrollment.
* Subject must be able to understand and give informed consent.

Exclusion Criteria:

* Age > 75 years old.
* Subject who is pregnant or breastfeeding or is unwilling to use adequate contraception.
* Subject who has had a previous chemotherapy for metastatic disease.
* Subject who has history of cardiac disease, with New York Heart Association Class II or greater with congestive heart failure.
* Subject who has clinically significant hepatic disease in regard to Hepatitis B, Hepatitis C, cirrhosis, or other liver diseases unrelated to the underlying metastatic breast cancer.
* Subject who has uncontrolled bacterial, viral, or fungal infection.
* Subject who exhibits confusion or disorientation.
* Subject with any condition which would prevent adequate follow-up.
* Subject who has received radiotherapy in the last 4 weeks.
* Subject with any other active primary tumor under treatment, except basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Subject who has brain metastasis.
* Subject who is not able to give informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to response; Duration of response; Time to progression; Survival | With complete or partial response, subjects will be re-evaluated 4 weeks later to confirm the initial observation; Follow-up for a minimum of one year for survival.

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF), (MUGA Scan); Radiological imaging; Examination of adverse events, laboratory data, vital signs | LVEF following cycles 2, 4, 5, and 6 of study drug; Radiological imaging every 6 weeks.

REFERENCES:
- [Result] Trudeau ME, Clemons MJ, Provencher L, Panasci L, Yelle L, Rayson D, Latreille J, Vandenberg T, Goel R, Zibdawi L, Rahim Y, Pouliot JF. Phase II multicenter trial of anthracycline rechallenge with pegylated liposomal doxorubicin plus cyclophosphamide for first-line therapy of metastatic breast cancer previously treated with adjuvant anthracyclines. J Clin Oncol. 2009 Dec 10;27(35):5906-10. doi: 10.1200/JCO.2009.22.7504. Epub 2009 Oct 26. PMID 19858391